CLINICAL TRIAL: NCT07251842
Title: Understanding the Metabolic Availability of Methionine in High Calcium Tempeh (TempeCalTM) Chips Among Reproductive-Age Women by Using the Stable Isotope Technique
Brief Title: Metabolic Availability of Methionine in Tempeh Chips Among Reproductive-age Women Using Indicator Amino Acid Oxidation (IAAO) Method
Acronym: IAAO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FRGS/1/2024/SKK06/UKM/02/3
Record Dates: First submitted 2025-11-17; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Healthy Women of Child Bearing Potential
Keywords: IAAO; Metabolic availability; tempeh
MeSH Terms: interventions — Eating

STUDY DESIGN:
Intervention Model Description: Each subject will randomly receive 4 levels of methionine provided as free amino acids, 3 levels of methionine provided as tempeh chips for a total of 7 studies x 3 days per study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- metabolic availability of methionine in tempeh chips (Experimental): Participants will undergo a pre-study assessment and will then complete up to seven experimental sessions over approximately 1.5-2 months.
  Each experimental set lasts 3 days. During the first 2 days (Adaptation Days), participants will consume four meals per day consisting of a protein liquid drink and protein-free cookies and/or tempeh chips provided by the investigators.
  Interventions: Other: dietary intakes; Other: Dietary intake

INTERVENTIONS:
Other: dietary intakes — Four levels of methionine intake provided via a crystalline amino acid mixture.
  Other Names: crystalline amino acid mixture
Other: Dietary intake — Three levels of methionine intake derived from tempeh chips.
  Other Names: tempeh chips

SUMMARY:
The goal of this study is to determine the protein quality of soybean tempeh in the form of chips. The main objective of this study is to determine how much methionine in tempeh can be used by reproductive-age women using the stable isotope method. The tempeh will be studied in the form of chips.

This research is being done to bridge the gap between the knowledge of protein requirements and the amount of food needed to meet those requirements. Results from this study will be important to confirm the protein quality of tempeh and thus provide a new alternative good protein source for humans, especially vegetarians and those with low socioeconomic status.

Each participant will undergo seven experimental trials randomly. During four experimental trials, methionine intake will be obtained from a crystalline amino acid mixture, and during another three experimental trials, it will be obtained from tempeh chips. Each experimental trial will take three days, consisting of two adaptation days and one study day. During the two adaptation days, four equal meals per day will be consumed by the participants at their own place. On the study day, participants will need to come to the research unit of the National University of Malaysia, Kuala Lumpur campus, to consume nine hourly meals. In addition, during the study day, participants will also need to have their breath samples collected, their expired carbon dioxide rate measured, and consume a stable isotope.

DETAILED DESCRIPTION:
For the pre-study assessment, participants will be required to measure their body weight, height, and resting energy expenditure (REE) using indirect calorimetry.

The study protocol is a 3-day experimental protocol consisting of 2 adaptation days and 1 indicator amino acid oxidation (IAAO) study day. For each 3-day experimental protocol, participants will be provided with either a reference diet for 3 days or a tempeh diet for 3 days. To begin another 3-day experimental protocol for the same participant, at least a 1-week interval will be required to ensure complete washout of the tracer.

During each adaptation period, every participant will be given 4 equal meals per day (breakfast, lunch, dinner, and snack) that fulfill 100% of their daily energy and protein requirements (Energy requirement = Resting Energy Expenditure (REE) × 1.7; Protein requirement = 1.0 g/kg/day × body weight). Meals provided will include a protein-free formula (required), protein-free butterscotch cookies (required), a crystalline amino acid mixture, or a combination of the crystalline amino acid mixture with tempeh chips. The meals should be finished by participants within 15 minutes. A daily multivitamin supplement and a 500 mg choline supplement will also be provided. In addition to plain water, only one cup of tea or coffee without sugar or cream is allowed during the adaptation days.

During the IAAO study period, after an overnight fast of 12 hours, participants will attend the metabolic laboratory at Kolej Tun Syed Nasir (KTSN) for 8 hours. A total of 9 isonitrogenous and isocaloric hourly meals will be provided, with each meal contributing 1/10 of the total energy requirement (REE × 1.5) and protein requirement (1.0 g/kg/day). Meals will consist of a protein-free formula (required), protein-free butterscotch cookies (required), and either a crystalline amino acid mixture or a combination of the crystalline amino acid mixture with tempeh chips. Each meal should be consumed within 15 minutes. The total meals provided will meet 90% of the participants' energy and protein requirements. During the experimental day, a daily multivitamin supplement and 500 mg of choline will also be provided.

During the first to fourth meals, participants will only be required to consume the provided meals. Starting from the fifth meal, participants will receive a constant oral isotope incorporation. Phenylalanine, an indispensable amino acid whose final metabolism produces carbon dioxide, will be used as the tracer to measure oxidation. In addition, NaH13CO3 (¹³C-sodium bicarbonate) will be administered as a priming dose to allow 13CO2(carbon-13 labeled CO₂) in the breath to reach a plateau within 2-3 hours. A dose of 0.176 mg/kg of NaH13CO3 and 0.66 mg/kg of L-[1-13C]phenylalanine will be given as the priming isotope during the fifth meal. From the fifth meal until the last meal, 1.2 mg/kg of L-[1-13C]phenylalanine will be provided continuously. The amount of phenylalanine provided as the tracer (excluding the priming isotope) will be subtracted from the dietary provision to maintain a total phenylalanine intake of 30 mg/kg/day. A total of 40 mg/kg/day (160% of the total aromatic amino acid requirement) of tyrosine will also be provided to ensure that no labeled phenylalanine is hydroxylated to meet the tyrosine requirement. After the fifth meal, the expired carbon dioxide production rate (VCO2) will be measured using indirect calorimetry for 15 minutes.

For breath sample collection, samples will be collected every 15 minutes before the tracer protocol is initiated (i.e., before the fifth meal) and every 15 minutes after isotopic steady state is reached (approximately 2.5 hours after isotope administration) until the end of the study. Additional breath samples will be collected 30 minutes after the end of the study. Each breath sample will be collected in triplicate using 10 mL non-silicon-coated tubes. The enrichment of 13CO2 in the breath will be analyzed using a continuous-flow isotope ratio mass spectrometer and expressed as atom percent excess (APE) over baseline. The fraction of 13CO2 (F13CO2) from L-[1-13C]phenylalanine oxidation relative to the amount administered will be calculated.

Using a linear mixed-effects regression model, the reference and test IAAO response slopes will be generated from F13CO2 measurements and their corresponding methionine intakes, with a common origin of the F13CO2 response at the base methionine intake. The metabolic availability (MA) of methionine in the test protein will be determined by the slope-ratio method using the following equation:

MA (%) = (Test protein / Reference protein) × 100.

ELIGIBILITY:
Inclusion Criteria:

* Universiti Kebangsaan Malaysia Kuala Lumpur campus female students and staffs aged 19 - 30 years old
* Malaysian
* Have consistent weight in the past 6 months
* Have a normal body fat percentage (20% - 29.9%)

Exclusion Criteria:

* Pregnant women
* Lactating women
* Reported serious medical or surgical ailments 3 months prior to start of the study
* On dietary or nutrient supplements or who had taken antibiotics 4 weeks before the initiation of the study
* Smoking
* Allergy to soybean
* Excessively high protein intake in the past 6 months

Ages: 19 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Metabolic availability of methionine in tempeh chips | From enrollment to the end of treatment at 8 weeks
  Using the Indicator Amino Acid Oxidation (IAAO) method to determine the MA of methionine in tempeh that is prepared in the chips form

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Kebangsaan Malaysia Kampus Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rafii M, Pencharz PB, Boileau K, Ball RO, Tomlinson C, Elango R, Courtney-Martin G. Metabolic Availability of Methionine Assessed Using Indicator Amino Acid Oxidation Method, Is Greater when Cooked Lentils and Steamed Rice Are Combined in the Diet of Healthy Young Men. J Nutr. 2022 Jun 9;152(6):1467-1475. doi: 10.1093/jn/nxac049. PMID 35218191